CLINICAL TRIAL: NCT06344494
Title: The Cardiac Intervention Imaging Clinical Trial of an Intracardiac Ultrasound Catheter and Ultrasound System
Brief Title: Cardiac Interventional ICE Imaging Trial
Acronym: INTELICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ICE Intelligent Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INTELICE-CTP-2401
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Structural Heart Diseases; Atrial Septal Defect; Patent Foramen Ovale; Arrhythmias, Cardiac; Atrial Fibrillation; Supraventricular Tachycardia; Valve Disease, Heart
Keywords: Intracardiac echocardiography
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent; Arrhythmias, Cardiac; Atrial Fibrillation; Tachycardia, Supraventricular; Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects will undergo planned intracardiac interventional procedures utilizing the Arch EchoTM Intracardiac Ultrasound catheter and combined ultrasound system.
  Interventions: Device: Arch EchoTM Intracardiac Ultrasound catheter and ultrasound system
- Control group (Active Comparator): Subjects will undergo planned intracardiac interventional procedures utilizing the SOUNDSTAR 3D Diagnostic Ultrasound catheter and ACUSON P500 system.
  Interventions: Device: SOUNDSTAR 3D Diagnostic Ultrasound catheter and ACUSON P500 system

INTERVENTIONS:
Device: Arch EchoTM Intracardiac Ultrasound catheter and ultrasound system — Novel ICE catheter and combined ultrasound system
  Arms: Experimental group
Device: SOUNDSTAR 3D Diagnostic Ultrasound catheter and ACUSON P500 system — Commercially available devices
  Arms: Control group

SUMMARY:
The INTELICE trial is a prospective, multicenter, 1:1 randomized controlled non-inferiority study. It aims to compare a novel intracardiac echography (ICE) catheter and combined ultrasound system with existing commercial ones. The evaluation will be conducted on patients undergoing planned intracardiac interventional process.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll adult patients undergoing cardiac interventions, who will be randomly assigned to either the experimental device group or the control group.

The main endpoint of the INTELICE trial is the image quality rate of intracardiac echocardiography, which will be evaluated by three experienced sonographers from the core laboratory, while the operator's image quality assessment serves as a secondary endpoint. In addition, secondary endpoints include clinical success rate, technical success rate, procedure time, and evaluation for the experimental devices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, ≤90 years, of any gender.
* Subjects deemed suitable for the utilization of ICE catheters during cardiac interventional procedures, as determined by investigators:

  1. Requirement for ICE imaging of the heart;
  2. Requirement for ICE imaging of great vessels;
  3. Requirement for ICE imaging of other intracardiac devices.
* Subjects themselves or their guardians must possess the ability to comprehend the purpose of this study, demonstrate adequate compliance with the protocol, and sign the informed consent form.

Exclusion Criteria:

* Anticipated vascular access (e.g., femoral vein, inferior vena cava, subclavian vein, internal jugular vein) cannot meet the procedure needs.
* PLT <100*109/L or INR >1.5.
* Intracardiac blood clots or severe peripheral vascular disease (e.g., deep vein thrombosis, aneurysm, atherosclerosis).
* Sepsis, pyemia, or severe systemic infection.
* NYHA Class IV.
* History of cardiac or related cardiac areas surgery within 6 months.
* Inability to tolerate post procedure oral anticoagulants or antiplatelet drugs.
* Inability to tolerate or cooperate with the procedure.
* Pregnant or lactating women, women with a positive pregnancy test result within 7 days before enrollment.
* Participation in other clinical trials of drugs, biological agents or devices within 3 months before screening.
* Other exclusive circumstances determined by the investigators, where the subject is deemed unsuitable for enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Image quality | Up to 6 months
  The image quality will be assessed by three cardiac sonographers. Sonographers will score based on image parameters such as image clarity, penetration, temporal and spatial resolution, blood flow, etc. The evaluation with utilize a 1-5 scale scoring system. A score of 5 indicates that the images are excellent and suitable for clinical needs, while a score of 4 suggests good quality. 3 indicates that the image has flaws but still meets the clinical needs. Scores of 1 and 2 signify poor or bad image quality, which can affect clinical diagnosis and treatment.

SECONDARY OUTCOMES:
Image quality | Up to 48 hours
  Adequate image quality will be assessed by the operators using the same evaluation criteria as the sonographers. However, the operator's responses are simplified and not encompass all different modes of ultrasound.
Procedure success | Up to 24 hours
  Interventional procedure success rate.
Technical success | Up to 24 hours
  Success delivery of ICE catheters to the target position. The operator aims to visualize a particular heart structure and requires the ICE catheter to be positioned at a specific site, such as the right atrium, right ventricular including outflow tract or left atrium, etc. The determination of whether the catheter has been successfully delivered to target locations is made by the operators.
Procedure time | Up to 24 hours
  The time from vascular puncture to completion.

OTHER OUTCOMES:
Device performance | Up to 24 hours
  Device performance evaluation by the investigator. The assessment will primarily focus on catheter parameters including deliverability, deflectability, compatibility, etc. A scoring system will be employed, where 5 points indicate the highest level of satisfaction, 3 points signify meeting the minimum requirements, and 1 or 2 points indicate dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Deyong Long, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Bejing
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The First Hospital Of Jilin University, Changchun, Jilin
  - Shanghai General Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No